CLINICAL TRIAL: NCT05980702
Title: Safety and Efficacy of Four Courses of Pembrolizumab Combined With Carboplatin and Albumin-binding Paclitaxel Versus Two Courses of Neoadjuvant Therapy in Patients With Resectable Head and Neck Squamous Cell Carcinoma (T3 or T4, N0) : An Optimal Efficacy Study (Prospective, Two-arm, Phase II)
Brief Title: 4 Courses vs 2 Courses of Pembrolizumab Combined With Carboplatin and Albumin-binding Paclitaxel of Neoadjuvant Therapy in HNSCC
Acronym: HNC-SYSU-002
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-219-02
Record Dates: First submitted 2023-06-05; First posted 2023-08-08 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: HNSCC; Oral Cancer; PD-1
Keywords: HNSCC; Oral Cancer; PD-1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 courses arm (Experimental): Drug:Pembrolizumab , Carboplatin,albumin-bound paclitaxel Patients receive Pembrolizumab IV on day 1, albumin-bound paclitaxel IV on day 1 and carboplatin IV on day 1 . Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Then surgery.
  Interventions: Drug: Pembrolizumab+Carboplatin+albumin-bound paclitaxel:4 courses
- 2 courses arm (Active Comparator): Drug:Pembrolizumab , Carboplatin,albumin-bound paclitaxel Patients receive Pembrolizumab IV on day 1, albumin-bound paclitaxel IV on day 1 and carboplatin IV on day 1 . Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Then surgery.
  Interventions: Drug: Pembrolizumab+Carboplatin+albumin-bound paclitaxel:2 courses

INTERVENTIONS:
Drug: Pembrolizumab+Carboplatin+albumin-bound paclitaxel:4 courses — Pembrolizumab,+Carboplatin+albumin-bound paclitaxel Pembrolizumab (IV), dose= 200mg , day=1 , cycle length: 21 days. Carboplatin (IV), dose=300mg/m2, day= 1, cycle length: 21 days. albumin-bound paclitaxel (IV), dose=260mg/m2, day= 1, cycle length: 21 days.
  Intervention: Drug: Pembrolizumab, Carboplatin, albumin-bound paclitaxel:4 cycles
  Arms: 4 courses arm
Drug: Pembrolizumab+Carboplatin+albumin-bound paclitaxel:2 courses — Pembrolizumab,+Carboplatin+albumin-bound paclitaxel Pembrolizumab (IV), dose= 200mg , day=1 , cycle length: 21 days. Carboplatin (IV), dose=300mg/m2, day= 1, cycle length: 21 days. albumin-bound paclitaxel (IV), dose=260mg/m2, day= 1, cycle length: 21 days.
  Intervention: Drug: Pembrolizumab , Carboplatin, albumin-bound paclitaxel:2 cycles
  Arms: 2 courses arm

SUMMARY:
In this study, 200 patients with resectable head and neck squamous cell carcinoma (T3 or T4, N0) were enrolled and preoperatively combined with pembrolizumab (PD-1 inhibitor), carboplatin, and albumin-binding paclitaxel. The subjects were randomly divided 1:1 into four treatments and two treatments. The imaging and pathological changes of tumor and paracancer tissues before and after treatment were observed. Clinical information, such as pathological grade, stage, treatment, prognosis, serology, imaging, etc., was collected to evaluate the safety and efficacy of 4-course pembrolizumab combined with carboplatin and albumin-binding paclitaxel compared with 2-course neoadjuvant therapy for resectable oral and oropharyngeal squamous cell carcinoma. This is a prospective, one-arm, phase II clinical study.

Main purpose By calculating pathological complete response (pCR) in the experimental group, we evaluated the efficacy (optimality) of four courses of pembrolizumab combined with carboplatin and albumin-binding paclitaxel compared with two courses of neoadjuvant therapy for resectable oral and oropharyngeal squamous cell carcinoma (T3 or T4, N0).

At the same time, this study evaluated the safety of medication, specifically: The severity of adverse events associated with neoadjuvant therapy will be graded according to NCI CTCAE (version 5.0) during this study and during follow-up, and the occurrence of adverse events in the experimental and control groups will be compared. To evaluate the safety of 4-course Pembrolizumab combined with carboplatin and albumin-binding paclitaxel compared with 2-course neoadjuvant therapy for resectable oral and oropharyngeal squamous cell carcinoma (T3 or T4, N0).

Secondary Purpose

1. The event-free survival (EFS) of the two groups were compared;
2. The main pathological response rate (MPR) of the two groups were compared;
3. pTR of the two groups was compared;
4. Overall survival (OS) of the two groups was compared;
5. The radiological responses of the two groups were compared;
6. The operation delay rate of the two groups was compared; Exploratory purpose For the response of enrolled patients after treatment, group treatment was conducted according to the guidelines, and stratified factors influencing the prognosis and treatment plan of immunotherapy were explored according to stratification. The stratification factors taken into consideration are: P16 status, smoking history, TNM stage, tumor reduction (MPR condition), presence of risk factors (according to the guidelines, risk factors are presence of episopercular invasion, positive incisal margin, proximal incisal margin, pT3 or pT4, pN2 or pN3 lymph nodes located in the IV and V regions of the neck, Nerve invasion, vascular invasion, etc.). The purpose of this study was to stratified risk factors for evaluating the efficacy of pembrolizumab combined with carboplatin and albumin-paclitaxel in neoadjuvant therapy for resectable head and neck squamous cell carcinoma. At the same time, hematological, pathological and fecal indicators collected in the design of the experiment were collected. Correlation analysis was conducted to statistically analyze the relationship between these indicators and the therapeutic effect of the program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age ≤65 years of age;
* cytological or histological diagnosis of surgically resectable head and neck squamous cell carcinoma with the following stages: T3 or T4, N0;
* According to the solid tumor efficacy evaluation criteria (RECIST version 1.1), there was at least one radiologically measurable lesion; First-line patients: have not previously received any systemic antitumor therapy for advanced/metastatic disease. Patients who had previously received platinum-containing adjuvant/neoadjuvant chemotherapy, or had received radical chemoradiotherapy for advanced disease, if the interval between disease progression or recurrence and the end of the last chemotherapy drug treatment was at least 6 months, were allowed to be enrolled in this study.
* ECOG score 0-1;
* Expected survival time > 3 months;
* Adequate organ function, subject shall meet the following laboratory indicators:

  1. The absolute value of neutrophil granulocyte (ANC) ≥1.5x109/L in the last 14 days without the use of granulocyte colony stimulating factor;
  2. Platelets ≥100×109/L without blood transfusion in the past 14 days;
  3. Hemoglobin &gt without blood transfusion or use of erythropoietin within the last 14 days; 9g/dL;
  4. Total bilirubin ≤1.5× upper limit of normal value (ULN);
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN in patients with liver metastasis);
  6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
  7. Good coagulation function, defined as International Standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. Subjects whose baseline TSH is outside the normal range can be enrolled if total T3 (or FT3) and FT4 are within the normal range;
  9. The myocardial enzyme profile was within the normal range (if the researchers comprehensively judged that the simple laboratory abnormality was not clinically significant, it was also allowed to be included);
  10. For female subjects of childbearing age, a urine or serum pregnancy test should be tested negative within 3 days prior to receiving the first study drug administration (day 1 of Cycle 1). If the urine pregnancy test results cannot be confirmed negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy;
  11. If there is a risk of conception, all subjects (male or female) shall use contraception with an annual failure rate of less than 1% for the entire duration of treatment up to 120 days after the last study drug administration (or 180 days after the last chemotherapeutic drug administration).

Exclusion Criteria:

* Malignant diseases other than head and neck squamous cell carcinoma diagnosed within 5 years prior to initial administration (excluding basal cell carcinoma of the skin after radical treatment, squamous epithelial carcinoma of the skin, and/or carcinoma in situ after radical excision);
* Currently participating in an interventional clinical study, or receiving other investigational drugs or using investigational devices within 4 weeks prior to initial dosing;
* Previous treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulus or synergistic inhibition of T cell receptors (e.g., CTLA-4, OX-40, CD137);
* Systemic treatment with Chinese patent drugs or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control pleural effusion) with indications of anti-head and neck squamous cell carcinoma within 2 weeks before the first administration;
* An active autoimmune immune disease requiring systemic treatment (e.g. with disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to initial administration. Alternative therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* Was receiving systemic glucocorticoid therapy (excluding nasal, inhalation, or other routes of topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days prior to initial administration; Note: Physiological doses of glucocorticoids (≤10 mg/ day of prednisone or equivalent) are permitted;
* Clinically uncontrollable pleural effusion/abdominal effusion (patients with no need to drain effusion or no significant increase of effusion after 3 days of stopping drainage could be included in the group);
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Those who are known to be allergic to the active ingredients or excipients of the drug in this study, Pabolizumab, carboplatin and albumin-binding paclitaxel;
* Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss);
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
* Untreated active hepatitis B (defined as HBsAg positive coupled with a detected HBV-DNA copy number greater than the upper limit of normal in the laboratory of the study center); Note: Hepatitis B subjects who meet the following criteria can also be enrolled:1) HBV viral load &lt before initial administration; At 1000 copies /ml (200 IU/ml), subjects should receive anti-HBV therapy to avoid viral reactivation throughout the study treatment period.2) For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required
* Active HCV infected subjects (HCV antibody positive and HCV-RNA level above the lower limit of detection);
* Received live vaccine within 30 days prior to initial administration (cycle 1, day 1); Note: Inactivated injectable virus vaccine against seasonal influenza is permitted for 30 days prior to initial administration; But live attenuated influenza vaccines administered intranasally are not allowed.
* Pregnant or lactating women;
* There is any serious or uncontrolled systemic disease, such as:

  1. The resting electrocardiogram (ECG) presents significant and severely uncontrollable abnormalities in rhythm, conduction or morphology, such as complete left bundle branch block, Ⅱ degree or above heart block, ventricular arrhythmia or atrial fibrillation;
  2. Unstable angina pectoris, congestive heart failure, and NYHA grade ≥ 2 chronic heart failure;
  3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before treatment;
  4. Poor blood pressure control (systolic > 140 mmHg, diastolic > 90 mmHg);
  5. A history of non-infectious pneumonia requiring glucocorticoid therapy or clinically active interstitial lung disease within 1 year prior to initial administration;
  6. Active pulmonary tuberculosis;
  7. There is an active or uncontrolled infection that requires systemic treatment;
  8. Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
  11. Urine routine indicated urine protein ≥++, and confirmed 24 hours urine protein quantity > 1.0 g;
  12. Patients with mental disorders and unable to cooperate with treatment;
* Medical history or evidence of disease that may interfere with test results, prevent participants from participating fully in the study, abnormal values of treatment or laboratory tests, or other conditions that the investigator considers unsuitable for enrollment. The Investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-04-03 (Estimated); Study Completion 2030-04-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events graded by CTCAE v5.0 | Time Frame: 90 days after surgery
  Percentage of adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0). Change From Baseline 90 days after surgery.
percentage of pathologic complete response(pCR) | 6 weeks
  The absence rate(Percentage) of invasive/in situ cancer and/or axillary lymph nodes.Change From Baseline from 6 weeks.

SECONDARY OUTCOMES:
Event-free survival (EFS) | 5 years
  In cancer, the length(measured by months) of time after primary treatment for a cancer ends that the patient remains free of certain complications or events that the treatment was intended to prevent or delay.
Overall survival(OS) | 5 years
  The time(measured by months) from day 1 of study treatment until death from any cause.
Operation delay rate | 2 months
  Rate(percentage) of patients with an Unplanned Delay to Surgery defined as any change to scheduled surgery date considered to be at least possibly related to neoadjuvant treatment.
Radiographic Response | 6 weeks
  Radiographic response to treatment as defined by RECIST 1.1. They are grouped by PR, CR,SD,PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No